CLINICAL TRIAL: NCT06037174
Title: Comparison of Quality of Life Between Patients with Early Differentiated Thyroid Cancer Undergoing Minimally Invasive and Open Surgery: a Prospective Cohort Study
Brief Title: Comparison of Quality of Life in Patients with Differentiated Thyroid Carcinoma Undergoing Different Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Xiaoming Huang, Professor; Director, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: SYSKY-2023-472-01
Record Dates: First submitted 2023-06-16; First posted 2023-09-14 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2023-12

CONDITIONS: Thyroid Cancer
Keywords: thyroid cancer; quality of life; minimally invasive; surgery
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Minimally Invasive Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — thyroid function test, thyroglobin, etc.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- minimally invasive surgery: undergoing thyroidectomy with endoscopy-assisted subclavian approach, robot-assisted transaxillary approach, robot-assisted transoral approach, robot-assisted retroauricular approach, etc.
  Interventions: Procedure: minimally invasive procedure
- traditional open surgery: undergoing thyroidectomy with tradition open surgery
  Interventions: Procedure: Conventional Open Surgery

INTERVENTIONS:
Procedure: minimally invasive procedure — different minimally invasive approach to complete thyroidectomy, including endoscopy-assisted subclavian approach, robot-assisted transaxillary or transoral approach (not leaving scar on the neck)
  Groups: minimally invasive surgery
Procedure: Conventional Open Surgery — Conventional Open Surgery
  Groups: traditional open surgery

SUMMARY:
The incidence of thyroid cancer has increased rapidly in recent years, especially in women. Early differentiated thyroid cancer has a good prognosis, and surgery is the main treatment. Traditional open surgery would leave a scar on the neck. However, emerging minimally invasive procedures can avoid the scar on the neck, resulting in better aesthetic effect, which would have an impact on the quality of life of patients to a certain degree.

This study intend to follow up patients regularly with early differentiated thyroid cancer undergoing different surgery. The quality of life, voice, scar would be assessed by authoritative questionaires or scales. We hope to demonstrate that minimally invasive surgery is better than traditional open surgery in order to provide reliable evidence for clinical practice.

DETAILED DESCRIPTION:
The incidence of thyroid cancer has increased rapidly in recent years, especially in women. Differentiated thyroid cancer takes the largest proportion in thyroid cancer, but it has a good prognosis. For early differentiated thyroid cancer, surgery is the main treatment. Traditional open surgery would leave a scar on the neck, which is especially troublesome for female patients. However, emerging minimally invasive procedures, such as endoscopy-assisted subclavian approach, robot-assisted transaxillary or transoral approach, etc., can avoid the scar on the neck, resulting in better aesthetic effect, which would have an impact on the quality of life of patients to a certain degree.

This study intend to follow up patients regularly with early differentiated thyroid cancer undergoing surgery according to a prospective cohort design. The evaluation questionnaires including quality of life, voice and scar would be completed to demonstrate that minimally invasive surgery is better than traditional open surgery not only in the way of effectiveness, but also in the quality of life. We hope to provide reliable evidence for clinical practice by this study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and < 70 years;
* Biopsy or surgical pathology indicated differentiated thyroid carcinoma (papillary thyroid carcinoma, follicular carcinoma);
* stage T1~T3a, N0~N1a, M0;
* Ability to read and write Chinese;
* Willingness to follow up.

Exclusion Criteria:

* Age < 18 years old or ≥70 years old;
* Biopsy or surgical pathology indicated medullary carcinoma or anaplastic thyroid carcinoma;
* Aggressive histology: tall cell, columnar cell, hobnail variant, etc.
* Mixed with medullary carcinoma or anaplastic thyroid carcinoma;
* High risk of recurrence (according to ATA guideline);
* Lateral cervical lymph node metastasis or distant metastasis;
* Suffer from other malignant tumors;
* History of thyroid surgery or cervical lymph node dissection;
* Cognition or behavior impairment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-10-10 (Estimated); Study Completion 2025-09-10 (Estimated)

PRIMARY OUTCOMES:
change of quality of life (SF-36) | baseline, 1month after surgery, 3 months after surgery, 6 months after surgery, 12 months after surgery
  change of the scores of the SF-36（36-item Short-Form）questionaire
change of quality of life (Thyca-Qol) | baseline, 1month after surgery, 3 months after surgery, 6 months after surgery, 12 months after surgery
  change of the scores of the Thyca-Qol（Thyroid Cancer-specific Quality of Life） questionaire

SECONDARY OUTCOMES:
voice handicap index | baseline, 1 month after surgery, 3 months after surgery, 6 months after surgery, 12 months after surgery
  assessment of quality of voice
scores of the surgical scar | 1 month after surgery, 3 months after surgery, 6 months after surgery, 12 months after surgery
  scores of the questionaires (POSAS) about scar
level of thyroglobulin | baseline, 1 month after surgery, 3 months after surgery, 6 months after surgery, 12 months after surgery
  an indicator to monitor tumor residual or recurrence
level of calcium | baseline, 1 month after surgery, 3 months after surgery, 6 months after surgery, 12 months after surgery
  to indicate whether the patient have hypocalcemia
operation duration | Intraoperative
  time for operation
blood loss | up to 1 week after surgery
  blood loss during operation
postoperative drainage | up to 1 week after surgery
  drainage volume after surgery
complications | baseline, 1 month after surgery, 3 months after surgery, 6 months after surgery, 12 months after surgery
  complication events after surgery, e.g. hoarseness, hypocalcemia, hemorrhage, seroma
satisfaction of the surgery | 1 month after surgery, 3 months after surgery, 6 months after surgery, 12 months after surgery
  Visual Analog Score for satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoming Huang, Study Director — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hopsital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No